CLINICAL TRIAL: NCT04100850
Title: Effectiveness of Aquatic Exercises for Improving Mental and Physical Health in Adults: Randomized Clinical Trial
Brief Title: Effectiveness of Aquatic Exercises for Improving Mental and Physical Health in Adults.
Acronym: AEforMH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal do vale do São Francisco (Other)
Responsible Party: Principal Investigator, Rodrigo Gustavo da Silva Carvalho, Principal Investigator, Universidade Federal do vale do São Francisco
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AE-Mental
Record Dates: First submitted 2019-09-20; First posted 2019-09-24 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Depression; Depressive Symptoms; Anxiety
Keywords: hydrotherapy; depression; anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Hydrotherapy

STUDY DESIGN:
Intervention Model Description: Watsu, Aquatic Exercises, Control
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aquatic Exercises (Experimental): Aquatic Exercises (AE) are water aerobics exercises and resistance exercises, classes will be supervised by a Physical Educator, in collective sessions of up to 30 people per class, twice a week, lasting 50 minutes, for two months.
  Interventions: Other: Aquatic Exercises
- Watsu (Active Comparator): The Watsu (water shiatsu) will be applied by a physical therapist, in individual sessions, twice a week, lasting 50 minutes, for two months in a warn pool (± 34°C). Watsu in particular prescribes transition of movements, once they are instituted, the therapist can create and adapt according to the limitations and restrictions that are encountered.
  Interventions: Other: Watsu
- Control (No Intervention): The control group will not receive any of these treatments (aquatic exercises and Watsu).

INTERVENTIONS:
Other: Aquatic Exercises — twice a week, lasting 50 minutes, for two months.
  Other Names: Aquatic Exercises (AE)
  Arms: Aquatic Exercises
Other: Watsu — twice a week, lasting 50 minutes, for two months.
  Other Names: Water Shiatsu (WS)
  Arms: Watsu

SUMMARY:
Objective: To compare the effectiveness between aquatic exercises (water aerobics versus Watsu) versus control groups, for improving the outcomes of depression, anxiety, stress, sleep quality, functionality, cognition and quality of life in patients with depression.

DETAILED DESCRIPTION:
Introduction: Considered as the "21st century disease", depression is a silent disease that stands out for its high prevalence and high morbidity, leading to serious consequences. With treatments made in aquatic environment, among them the Water aerobics and Watsu. Objective: To compare the effectiveness between aquatic exercises versus Watsu and versus control group, for improving the outcomes of depression, anxiety, stress, sleep quality, functionality, cognition and quality of life in patients with depression. Methods: This study will be a randomized clinical trial, which will last for two months with a follow-up of one month. All participants will be assessed using specific questionnaires for each outcome and an Improvement Perception Scale (MS). Seventy eight (78) patients with a medical diagnosis of depression, aged 18 to 60 years, who will be allocated to three groups (26 patients for each group) will be treated. GROUP 1: Aquatic exercises (aerobic and resistance), collective session, twice a week lasting 50 min; GROUP 2: Watsu (water shiatsu), individual session, twice a week lasting 50 min; Group 3: control, people with depression. Statistical analysis: Normality distribution will be by Shapiro-Wilk test. For comparisons of the means between and within the outcome groups will be used through Generalized Estimation Equations, with its own syntax, linear distribution and, when necessary, multiple comparisons will be performed using the Bonferroni test to identify differences. Will be calculated for comparisons between the final and initial moments and initial follow-up in each group, statistics such as: mean difference (95% CI), standard deviation of the difference, effect size (Cohen's d). The statistical significance adopted was 5% and the analyzes were performed using the statistical programs SPSS 22.0 and R 3.2.4. The intention-to-treat analysis will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60 years old;
* Sedentary and who have not had physical therapy and physical activity in the last three months;
* Clinical and cognitive conditions for performing pool activities and moderate aerobic exercise;
* Who have not undergone high complexity surgical procedures in the last six months; no neuro-musculosqueletal diseases;
* No contraindications to exercise; such as: urinary and / or fecal incontinence and dermatological diseases;
* Individuals with a medical diagnosis of depression.

Exclusion Criteria:

* If they have up to three absences during the intervention period;
* If they have any adverse effects, such as: allergy or dermatitis;
* Unable to continue study due to change of address or hospitalization.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 78 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Depression | change depression at 8 weeks and follow-up at 12 weeks
  Beck Depression Inventory (better 0-63 worse points)
Anxiety | change anxiety at 8 weeks and follow-up at 12 weeks
  Beck Anxiety Inventory (better 0-63 worse points)

SECONDARY OUTCOMES:
Stress | change stress at 8 weeks and follow-up at 12 weeks
  Depression, Anxiety and Stress Scale (DASS-21) (better 0 - worse >34)
Quality of Life Questionnaire | change quality of live at 8 weeks and follow-up at 12 weeks
  12-Item Short-Form Health Survey (SF-12) (worse 0 - better 100)
Sleep Quality | change sleep quality at 8 weeks and follow-up at 12 weeks
  Pittsburgh Sleep Quality Index (PSQI) (better 0 - worse 21)
Life Style Scale | change life style at 8 weeks and follow-up at 12 weeks
  Fantastic Life Style Scale (worse 0 - better 100)
Cognitive | change cognitive at 8 weeks and follow-up at 12 weeks
  Montreal Cognitive Assessment (MOCA) (worse 0 - better 30)
Functionally | change functionally at 8 weeks and follow-up at 12 weeks
  Six-minute Walk Test (6m-WT)

OTHER OUTCOMES:
Improvement Perception | pos (8 week)
  Improvement Perception Scale (0-7)

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo GS Carvalho, PhD, Principal Investigator — Physical Education College / UNIVASF
Locations (1):
- Physical Education College, Petrolina, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: No
Study Protocol, Randomized Clinical Trial